CLINICAL TRIAL: NCT00462917
Title: Risk Evaluation and Education for Alzheimer's Disease
Brief Title: REVEAL III: Risk Evaluation and Education for Alzheimer's Disease
Acronym: REVEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Robert C. Green, MD, MPH, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: IA0113; R01HG002213 (NIH)
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer Disease
Keywords: disease /disorder proneness /risk; family genetics; genetic counseling; genetic marker; genetic polymorphism; genetic screening; genetic susceptibility
MeSH Terms: conditions — Alzheimer Disease; Disease Susceptibility; Genetic Predisposition to Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pleiotropic info, in-person disclosure (Experimental): Incidental pleiotropic risk information, in addition to AD risk information, is disclosed in-person during an APOE-based genetic risk assessment
  Interventions: Behavioral: Pleiotropic info, in-person disclosure
- AD-only info, phone disclosure (Experimental): Alzheimer's disease risk information only is disclosed via telephone during an APOE-based genetic risk assessment
  Interventions: Behavioral: AD-only info, phone disclosure
- Pleiotropic info, phone disclosure (Experimental): Incidental pleiotropic risk information, in addition to AD risk information, is disclosed via telephone during an APOE-based genetic risk assessment
  Interventions: Behavioral: Pleiotropic info, phone disclosure
- AD-only info, in-person disclosure (Active Comparator): Alzheimer's disease risk information only is disclosed in-person during an APOE-based genetic risk assessment
  Interventions: Behavioral: AD-only info, in-person disclosure

INTERVENTIONS:
Behavioral: Pleiotropic info, in-person disclosure — Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping as well as additional pleiotropic information.
  Genetic counselors communicate results to participants during an in-person disclosure session.
  Arms: Pleiotropic info, in-person disclosure
Behavioral: AD-only info, in-person disclosure — Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping.
  Genetic counselors communicate results to participants during an in-person disclosure session.
  Arms: AD-only info, in-person disclosure
Behavioral: Pleiotropic info, phone disclosure — Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping as well as additional pleiotropic information.
  Genetic counselors communicate results to participants during a telephone disclosure session.
  Arms: Pleiotropic info, phone disclosure
Behavioral: AD-only info, phone disclosure — Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping.
  Genetic counselors communicate results to participants during an in-person disclosure session.
  Arms: AD-only info, phone disclosure

SUMMARY:
The purpose of this study is to provide healthy adults with genetic testing and information about their chances of developing Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease is a common condition affecting memory and thinking. Genes can sometimes be used to provide risk estimates for the eventual development of certain common diseases. Apolipoprotein E (APOE) is one gene that has been identified which can provide information about a person's chances of developing Alzheimer's diseases. Previous research explored the behavioral and psychological impact of receiving genetic risk information for Alzheimer's disease (AD). The REVEAL I Study, funded in 1999, showed that an Alzheimer's disease genetic risk assessment can be given to relatives of people with AD in a safe way. REVEAL II, which was funded in 2003, demonstrated that this same information can be given in a condensed education and counseling protocol without causing severe psychological harm. REVEAL III will further study different ways of providing genetic risk information for Alzheimer's disease.

Participation in this study will entail an initial screening phone call to determine eligibility, followed by a phone interview which will ask about demographic information and thoughts and feelings about AD. Participants will complete a mailed survey. Following completion of the survey, a genetic counselor will meet with the participant at the clinic to review family and medical history, administer additional questionnaires asking about AD and genetic testing, and draw blood for genetic testing. Results will be disclosed either in person or over the phone about 3 to 4 weeks later. The genetic counselor will make a brief follow-up phone call 1 week after that. The participant will visit the clinic twice to provide additional information, at 6 weeks and 6 months after disclosure. Finally, the participant will complete a mailed 12 month survey, and the genetic counselor will make a brief follow-up phone call.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years to 85 years old

Exclusion Criteria:

* Unable to visit a study site
* Current untreated depression or anxiety
* Family history of AD diagnosed under age 60
* More than one first-degree relative diagnosed with AD (e.g. Mother and brother)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Green, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (4):
- United States (4):
  - Howard University, Washington D.C., District of Columbia
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Background] Hipps YG, Roberts JS, Farrer LA, Green RC. Differences between African Americans and Whites in their attitudes toward genetic testing for Alzheimer's disease. Genet Test. 2003 Spring;7(1):39-44. doi: 10.1089/109065703321560921. PMID 12820701
- [Background] Roberts JS, LaRusse SA, Katzen H, Whitehouse PJ, Barber M, Post SG, Relkin N, Quaid K, Pietrzak RH, Cupples LA, Farrer LA, Brown T, Green RC. Reasons for seeking genetic susceptibility testing among first-degree relatives of people with Alzheimer disease. Alzheimer Dis Assoc Disord. 2003 Apr-Jun;17(2):86-93. doi: 10.1097/00002093-200304000-00006. PMID 12794385
- [Background] Roberts JS, Barber M, Brown TM, Cupples LA, Farrer LA, LaRusse SA, Post SG, Quaid KA, Ravdin LD, Relkin NR, Sadovnick AD, Whitehouse PJ, Woodard JL, Green RC. Who seeks genetic susceptibility testing for Alzheimer's disease? Findings from a multisite, randomized clinical trial. Genet Med. 2004 Jul-Aug;6(4):197-203. doi: 10.1097/01.gim.0000132688.55591.77. PMID 15266207
- [Background] LaRusse S, Roberts JS, Marteau TM, Katzen H, Linnenbringer EL, Barber M, Whitehouse P, Quaid K, Brown T, Green RC, Relkin NR. Genetic susceptibility testing versus family history-based risk assessment: Impact on perceived risk of Alzheimer disease. Genet Med. 2005 Jan;7(1):48-53. doi: 10.1097/01.gim.0000151157.13716.6c. PMID 15654228
- [Background] Roberts JS, Cupples LA, Relkin NR, Whitehouse PJ, Green RC; REVEAL (Risk Evaluation and Education for Alzheimer's Disease) Study Group. Genetic risk assessment for adult children of people with Alzheimer's disease: the Risk Evaluation and Education for Alzheimer's Disease (REVEAL) study. J Geriatr Psychiatry Neurol. 2005 Dec;18(4):250-5. doi: 10.1177/0891988705281883. PMID 16306249
- [Background] Roberts JS, Christensen KD, Green RC. Using Alzheimer's disease as a model for genetic risk disclosure: implications for personal genomics. Clin Genet. 2011 Nov;80(5):407-14. doi: 10.1111/j.1399-0004.2011.01739.x. Epub 2011 Jul 18. PMID 21696382
- [Result] Christensen KD, Uhlmann WR, Roberts JS, Linnenbringer E, Whitehouse PJ, Royal CDM, Obisesan TO, Cupples LA, Butson MB, Fasaye GA, Hiraki S, Chen CA, Siebert U, Cook-Deegan R, Green RC. A randomized controlled trial of disclosing genetic risk information for Alzheimer disease via telephone. Genet Med. 2018 Jan;20(1):132-141. doi: 10.1038/gim.2017.103. Epub 2017 Jul 20. PMID 28726810
- [Result] Christensen KD, Roberts JS, Whitehouse PJ, Royal CD, Obisesan TO, Cupples LA, Vernarelli JA, Bhatt DL, Linnenbringer E, Butson MB, Fasaye GA, Uhlmann WR, Hiraki S, Wang N, Cook-Deegan R, Green RC; REVEAL Study Group*. Disclosing Pleiotropic Effects During Genetic Risk Assessment for Alzheimer Disease: A Randomized Trial. Ann Intern Med. 2016 Feb 2;164(3):155-63. doi: 10.7326/M15-0187. Epub 2016 Jan 26. PMID 26810768
- [Result] Christensen KD, Roberts JS, Zikmund-Fisher BJ, Kardia SL, McBride CM, Linnenbringer E, Green RC; REVEAL Study Group. Associations between self-referral and health behavior responses to genetic risk information. Genome Med. 2015 Jan 31;7(1):10. doi: 10.1186/s13073-014-0124-0. eCollection 2015. PMID 25642295
- [Result] Besser AG, Sanderson SC, Roberts JS, Chen CA, Christensen KD, Lautenbach DM, Cupples LA, Green RC. Factors affecting recall of different types of personal genetic information about Alzheimer's disease risk: the REVEAL study. Public Health Genomics. 2015;18(2):78-86. doi: 10.1159/000368888. Epub 2015 Jan 24. PMID 25634646
- See also: Primary REVEAL Study web site (http://www.genomes2people.org/reveal/) — http://www.genomes2people.org/reveal/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pleiotropic Info, In-person Disclosure: Incidental pleiotropic risk information, in addition to Alzheimer's disease risk information, is disclosed in-person during an APOE-based genetic risk assessment
  Pleiotropic info, in-person disclosure: Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping as well as additional pleiotropic information.
  Genetic counselors communicate results to participants during an in-person disclosure session.
- AD-only Info, Phone Disclosure: Alzheimer's disease risk information only is disclosed via telephone during an APOE-based genetic risk assessment
  AD-only info, phone disclosure: Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping.
  Genetic counselors communicate results to participants during an in-person disclosure session.
- Pleiotropic Info, Phone Disclosure: Incidental pleiotropic risk information, in addition to Alzheimer's disease risk information, is disclosed via telephone during an APOE-based genetic risk assessment
  Pleiotropic info, phone disclosure: Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping as well as additional pleiotropic information.
  Genetic counselors communicate results to participants during a telephone disclosure session.
- AD-only Info, In-person Disclosure: Alzheimer's disease risk information only is disclosed in-person during an APOE-based genetic risk assessment
  AD-only info, in-person disclosure: Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping.
  Genetic counselors communicate results to participants during an in-person disclosure session.
Period: Overall Study
Arm/Group | Pleiotropic Info, In-person Disclosure | AD-only Info, Phone Disclosure | Pleiotropic Info, Phone Disclosure | AD-only Info, In-person Disclosure
Started | 72 | 75 | 66 | 77
Met With Genetic Counselor | 66 | 71 | 56 | 71
Received Risk Information | 64 | 70 | 55 | 68
Completed 6 Week Follow-up | 63 | 70 | 55 | 68
Completed 6 Month Follow-up | 63 | 68 | 55 | 66
Completed | 62 | 65 | 54 | 66
Not Completed | 10 | 10 | 12 | 11

BASELINE CHARACTERISTICS:
Population: Baseline population includes all participants who received genetic risk information, regardless of whether they completed follow-up time surveys.
Groups:
- Pleiotropic Info, In-person Disclosure: Incidental pleiotropic risk information, in addition to AD risk information, is disclosed in-person during an APOE-based genetic risk assessment
  Pleiotropic info, in-person disclosure: Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping as well as additional pleiotropic information.
  Genetic counselors communicate results to participants during an in-person disclosure session.
- Pleiotropic Info, Phone Disclosure: Incidental pleiotropic risk information, in addition to AD risk information, is disclosed via telephone during an APOE-based genetic risk assessment
  Pleiotropic info, phone disclosure: Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease based on APOE genotyping as well as additional pleiotropic information.
  Genetic counselors communicate results to participants during a telephone disclosure session.
- Total: Total of all reporting groups
Arm/Group | Pleiotropic Info, In-person Disclosure | AD-only Info, Phone Disclosure | Pleiotropic Info, Phone Disclosure | AD-only Info, In-person Disclosure | Total
Number analyzed (Participants) | 64 | 70 | 55 | 68 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12) | 57 (13) | 59 (13) | 59 (12) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 29 | 37 | 141
  Male | 28 | 31 | 26 | 31 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 13 | 4 | 16 | 38
  White | 59 | 55 | 50 | 51 | 215
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 64 | 70 | 55 | 68 | 257
Anxiety (Beck Anxiety Index: BAI) [Mean (Standard Deviation); unit: units on a scale] — Scores on the Beck Anxiety Index (BAI), a 21-item scale measuring general anxiety. Scores range from 0-63, with higher scores indicating greater anxiety.
  units on a scale | 2.7 (2.9) | 3.6 (3.4) | 3.8 (3.7) | 4.0 (3.8) | 3.5 (3.5)
Depression (Center for Epidemiological Studies Depression Scale: CES-D) [Mean (Standard Deviation); unit: units on a scale] — Scores on the Center for Epidemiological Studies Depression Scale (CES-D), a 20-item scale measuring general depression. Scores range from 0-60, with higher scores indicating greater general depression.
  units on a scale | 5.1 (4.6) | 5.5 (5.4) | 5.5 (5.0) | 6.6 (5.3) | 5.7 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiological Studies-Depression Scale (CES-D)
Description: A 20-item scale measuring general depression. Scores range from 0-60, with higher scores indicating greater general depression.
Time Frame: 6 weeks, 6 months, and 12 months post-disclosure
Population: "Number of participants analyzed" are the number of participants who received genetic risk information and completed the 6-week follow-up (256). At 6 months, 252 participants provided data. At 12 months, 247 participants provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pleiotropic Info, In-person Disclosure | AD-only Info, Phone Disclosure | Pleiotropic Info, Phone Disclosure | AD-only Info, In-person Disclosure
Number analyzed (Participants) | 63 | 70 | 55 | 68
score on a scale
  6 Weeks | 4.8 (5.0) | 7.0 (8.4) | 6.4 (6.4) | 5.5 (5.4)
  6 Months: number analyzed (Participants) | 63 | 68 | 55 | 66
  6 Months | 5.5 (7.0) | 6.6 (6.7) | 5.8 (6.4) | 6.1 (6.6)
  12 Months: number analyzed (Participants) | 62 | 65 | 54 | 66
  12 Months | 7.1 (8.2) | 7.6 (9.0) | 7.1 (7.0) | 6.2 (6.9)

2. Primary Outcome: Beck Anxiety Inventory (BAI)
Description: A 21-item scale measuring general anxiety. Scores range from 0-63, with higher scores indicating greater anxiety.
Time Frame: 6 weeks, 6 months, 12 months post-disclosure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pleiotropic Info, In-person Disclosure | AD-only Info, Phone Disclosure | Pleiotropic Info, Phone Disclosure | AD-only Info, In-person Disclosure
Number analyzed (Participants) | 63 | 70 | 55 | 68
score on a scale
  6 Weeks | 2.9 (3.6) | 4.1 (5.4) | 3.2 (4.2) | 3.1 (3.3)
  6 Months: number analyzed (Participants) | 63 | 68 | 55 | 66
  6 Months | 3.4 (5.4) | 3.4 (4.3) | 3.3 (3.8) | 3.0 (5.0)
  12 Months: number analyzed (Participants) | 62 | 65 | 54 | 66
  12 Months | 3.4 (5.5) | 4.0 (5.3) | 3.5 (3.4) | 3.8 (4.8)

3. Secondary Outcome: Impact of Events Scale (IES)
Description: A 15-item scale measuring distress specific to the test results received. Scores range from 0-75, with higher scores indicating greater test-related distress.
Time Frame: 6 weeks, 6 months, 12 months post-disclosure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pleiotropic Info, In-person Disclosure | AD-only Info, Phone Disclosure | Pleiotropic Info, Phone Disclosure | AD-only Info, In-person Disclosure
Number analyzed (Participants) | 63 | 70 | 55 | 68
score on a scale
  6 Weeks | 3.4 (6.4) | 4.5 (7.9) | 3.7 (6.3) | 3.8 (7.7)
  6 Months: number analyzed (Participants) | 63 | 68 | 55 | 66
  6 Months | 3.5 (8.7) | 4.0 (8.2) | 3.0 (4.2) | 3.2 (5.8)
  12 Months: number analyzed (Participants) | 62 | 65 | 54 | 66
  12 Months | 2.4 (5.9) | 4.0 (10.4) | 2.5 (5.2) | 3.3 (7.4)

ADVERSE EVENTS:
Arm/Group | Pleiotropic Info, In-person Disclosure | AD-only Info, Phone Disclosure | Pleiotropic Info, Phone Disclosure | AD-only Info, In-person Disclosure
Serious Adverse Events (participants affected / at risk) | 1/64 | 0/70 | 0/55 | 0/68
Other Adverse Events (participants affected / at risk) | 8/64 | 9/70 | 4/55 | 5/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pleiotropic Info, In-person Disclosure (N=64) | AD-only Info, Phone Disclosure (N=70) | Pleiotropic Info, Phone Disclosure (N=55) | AD-only Info, In-person Disclosure (N=68)
Death (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pleiotropic Info, In-person Disclosure (N=64) | AD-only Info, Phone Disclosure (N=70) | Pleiotropic Info, Phone Disclosure (N=55) | AD-only Info, In-person Disclosure (N=68)
Potential mood disorder (Psychiatric disorders) | 5 (5) | 8 (8) | 4 (6) | 5 (5) — BAI or CES-D scores above standard cutoffs for severe anxiety or depression, respectively; or increases of at least 15 points from baseline on BAI or CES-D scores at any follow up. Events are noted regardless of whether they are study-related
Hospitalization (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) — Participant was hospitalized. Events are reported regardless of whether they are study-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes